CLINICAL TRIAL: NCT05254197
Title: The Risk of Growth in Patients With Non-malignant Brain Tumor: SeOuL cOhort of Brain Tumor MONitoring (SOLOMON) Study
Brief Title: SeOuL cOhort of Brain Tumor MONitoring Study (SOLOMON)
Acronym: SOLOMON
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Chul-Kee Park, Professor, Seoul National University Hospital
Other Study IDs: SNUH-BTR01
Record Dates: First submitted 2022-02-14; First posted 2022-02-24 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Brain Tumor, Primary; Meningioma; Schwannoma; Pituitary Adenoma; Gliomas Benign
Keywords: Non-malignant brain tumor; Benign brain tumor; Meningioma; Schwannoma; Pituitary adenoma; Benign glioma
MeSH Terms: conditions — Brain Neoplasms; Meningioma; Neurilemmoma; Pituitary Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Retrospective cohort: The registry of this study was subjected to patients who were radiologically diagnosed with a non-malignant brain tumor at Seoul National University Hospital since 1998, and who have had MR re-examination after first MR exam because it was determined that immediate treatment would not be needed at the first visit to the hospital. Non-malignant brain tumors are defined as radiologically diagnosed primary intracranial neoplasms of CNS WHO grade 2 or lower and include meningioma, schwannoma, pituitary adenoma, and glioma suspected to be non-malignant. It is practically impossible to obtain informed consent from patients of this retrospective cohort, and consent was waived by the Institutional Review Board. Target population of this retrospective cohort is 1,500 tumors.
- Prospective cohort: The registry of this study was subjected to patients who were radiologically diagnosed with a non-malignant brain tumor at Seoul National University Hospital since February 2022, and who have had MR re-examination after first MR exam or will be re-examined because it was determined that immediate treatment would not be needed at the first visit to the hospital. Non-malignant brain tumors are defined as radiologically diagnosed primary intracranial neoplasms of CNS WHO grade 2 or lower and include meningioma, schwannoma, pituitary adenoma, and glioma suspected to be non-malignant. The cohort will consists of patients who agree to participate with written consent. Target population of this prospective cohort is 1,500 tumors.

SUMMARY:
The registry of this study was subjected to patients who were radiologically diagnosed with a non-malignant brain tumor at Seoul National University Hospital since 2001, and who have had magnetic resonance (MR) re-examination after first MR exam or will be re-examined because it was determined that immediate treatment would not be needed at the first visit to the hospital. In all MRs taken by patients, the date of imaging and the volume of the tumor are measured, and we aim to establish a natural growth history for non-malignant brain tumors.

DETAILED DESCRIPTION:
Non-malignant central nervous system (CNS) tumor accounts for 70% of all primary CNS tumors, and over 300,000 patients were diagnosed with non-malignant CNS tumor per year in the United States. Not much is known about the natural history of non-malignant CNS tumors, as it is often treated immediately upon detection. However, some of them, especially small and asymptomatic non-malignant CNS tumors should not be treated immediately upon diagnosis but are observed and followed-up by repeated magnetic resonance imaging (MRI). This study aims to make a prospective cohort of non-malignant CNS tumors that do not require immediate treatment and to quantitatively analyze which factors are related to the growth of tumors.

The registry of this study was subjected to patients who were radiologically diagnosed with a non-malignant brain tumor at Seoul National University Hospital since 2001, and who have had MR re-examination after first MR exam or will be re-examined because it was determined that immediate treatment would not be needed at the first visit to the hospital. Non-malignant brain tumors are defined as radiologically diagnosed neoplasms of CNS WHO grade 2 or lower among primary intracranial tumors and include meningioma, schwannoma, pituitary adenoma, and glioma suspected to be non-malignant.

ELIGIBILITY:
Inclusion Criteria for retrospective cohort

* Patients with radiologically diagnosed brain neoplasm of CNS WHO grade 2 or less since 1998
* Asymptomatic at first visit to the hospital
* Patients who, based on the up-to-date knowledge, did not necessarily require immediate treatment at the first hospital visit
* Patients who have had two or more MRs at least 3 months apart
* No previous radiotherapy or radiosurgery for the brain lesion
* 18 years old or more

Inclusion Criteria for prospective cohort

* Patients with newly diagnosed brain neoplasm of CNS WHO grade 2 or less
* Asymptomatic at first visit to the hospital
* Patients who, based on the up-to-date knowledge, did not necessarily require immediate treatment at the first hospital visit and who are going to take follow-up MR exams
* No previous radiotherapy or radiosurgery for the brain lesion
* 18 years old or more
* Patients who agree to participate by written consent

Exclusion Criteria

* Patients who lost follow-up before the second MR exam
* Patients requiring immediate treatment due to worsening of symptoms within 3 months of the first MR exam
* Patients suspected to have other than a neoplasm at follow-up MR exams

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Investigators defined the cohort population as adults with radiologically diagnosed non-malignant brain tumor that do not require immediate treatment who agree to participate.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor volume in each MRI | within 15 years after enrollment
  Measured tumor volume in each MRI
T2 signal intensity of tumor in each MRI | within 15 years after enrollment
  T2 signal intensity of tumor as a ratio to contralateral white matter

SECONDARY OUTCOMES:
Growth rate of tumor volume between MR exams (absolute volume) | within 15 years after enrollment
  Tumor volume changed on average per year
Growth rate of tumor volume between MR exams (volume ratio) | within 15 years after enrollment
  Percentage of tumors that change on average per year
Number of patients who eventually received treatment | within 15 years after enrollment
  Number of patients who eventually received treatment, such as surgery, radiosurgery, radiotherapy, or hormonal therapy.
Pre-treatment follow-up period for patients who eventually received treatment | within 15 years after enrollment
  Pre-treatment follow-up period for patients who eventually received treatment, such as surgery, radiosurgery, radiotherapy, or hormonal therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Kee Park, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
We have no plan to share our individual participant data because is is not permitted by the Institutional Review Board.

REFERENCES:
- [Result] Kim JH, Dho YS, Kim YH, Lee JH, Lee JH, Hong AR, Shin CS. Developing an optimal follow-up strategy based on the natural history of nonfunctioning pituitary adenomas. J Neurosurg. 2018 Sep 14;131(2):500-506. doi: 10.3171/2018.4.JNS172148. Print 2019 Aug 1. PMID 30215565
- [Result] Behbahani M, Skeie GO, Eide GE, Hausken A, Lund-Johansen M, Skeie BS. A prospective study of the natural history of incidental meningioma-Hold your horses! Neurooncol Pract. 2019 Dec;6(6):438-450. doi: 10.1093/nop/npz011. Epub 2019 Apr 17. PMID 31832214
- [Result] Reznitsky M, Petersen MMBS, West N, Stangerup SE, Caye-Thomasen P. The natural history of vestibular schwannoma growth-prospective 40-year data from an unselected national cohort. Neuro Oncol. 2021 May 5;23(5):827-836. doi: 10.1093/neuonc/noaa230. PMID 33068429